CLINICAL TRIAL: NCT06642129
Title: A Prospective Observational Study of Perioperative Lumbar Puncture Pressure and Shunt Valve Pressure Management in Patients with Traffic Hydrocephalus Undergoing Lumbopeitoneal Shunt Surgery
Brief Title: A Prospective Observational Study of Perioperative Lumbar Puncture Pressure and Shunt Valve Pressure Management in Patients with Communicating Hydrocephalus Undergoing Lumboperitoneal Shunt Surgery
Acronym: LPP-LPS
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Junfeng Feng, Chief Director of Brain Injury Center, RenJi Hospital
Other Study IDs: LY2024-070-B
Record Dates: First submitted 2024-09-15; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Hydrocephalus, Communicating
MeSH Terms: conditions — Hydrocephalus | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Oberservation Group: Patient requiring surgical treatment with lumboperitoneal shunt for communicating hydrocephalus
  Interventions: Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines

INTERVENTIONS:
Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines — Lumboperitoneal shunt (LPS) involves connecting the subarachnoid space of the lumbar spine to the peritoneal cavity through a pressure-adjustable unidirectional valve to shunt the appropriate amount of cerebrospinal fluid from the ventricles to the peritoneal cavity via the spinal canal, where it is absorbed through the peritoneum, to alleviate the increased intracranial pressure caused by the communicating hydrocephalus and the corresponding clinical symptoms.

SUMMARY:
Target population: patients 18 years of age or older who require surgical treatment with lumboperitoneal shunt surgery for traffic hydrocephalus Estimated sample size: 30 cases. Study design: this study is a multicenter prospective observational study, with lumbar puncture pressure measurement before and during surgery, and shunt valve setting pressure set according to the requirements of clinical practice in the hospital where it is performed, and the collection of relevant data, including preoperative lumbar puncture pressure, intraoperative lumbar puncture pressure after anesthesia, shunt valve initial pressure, shunt valve pressure at 6 months pressure, length of the intravertebral shunt, and length of the intraperitoneal shunt. Complications, shunt effects, and the number of shunt valve adjustments during the 6-month period were also observed and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or older;
2. Confirmed diagnosis of communicating hydrocephalus;
3. Signed informed consent for surgery and informed consent for research.

Exclusion Criteria:

1. Pregnant women;
2. Inappropriate for lumboperitoneal shunt surgery despite the diagnosis of communicating hydrocephalus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age and older who require surgical treatment with lumboperitoneal shunt for communicating hydrocephalus
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
primary outcome | preoperation to 6 months after surgery
  1. Measurement of preoperative bedside lumbar puncture pressure(cmH2O);
  2. Measurement of lumbar puncture pressure after anesthesia during lumboperitoneal shunt surgery(cmH2O) ;
  3. Initial setting of shunt valve;
  4. Setting of shunt valve at 6 months after lumboperitoneal shunt surgery

SECONDARY OUTCOMES:
secondary outcome | preoperation to 6 months after surgery
  The numbers of complications related to the lumboperitoneal shunt at 6 months after the shunt operation, including: subdural hemorrhage, ventricular hemorrhage, intracerebral hemorrhage, subdural effusion, shunt obstruction, resetting the shunt, intracranial infection, and epilepsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided